CLINICAL TRIAL: NCT06552676
Title: Risk Factors for Neck Phlegmon After Percutaneous Tracheostomy in ICU
Acronym: SORCERER
Status: Recruiting | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: SORCERER - 24088
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Tracheostomy Complication; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Percutaneous tracheostomy: Patients receiving percutaneous tracheostomy for any reason during their ICU stay
  Interventions: Procedure: Percutaneous tracheostomy

INTERVENTIONS:
Procedure: Percutaneous tracheostomy — Percutaneous tracheostomy is a widely used technique in intensive care. It involves creating a passage between the tracheal lumen and the outside, through which a cannula is placed.

SUMMARY:
Primary Purpose: To investigate the incidence and risk factors related to the appearance of tracheal phlegmon in patients undergoing percutaneous tracheostomy.

Participant Population/Primary Condition: Patients admitted to Intensive Care

Main Questions Aims to Answer:

1. - What are the risk factors associated with the development of tracheal phlegmon percutaneous tracheostomy?
2. - How does the appearance of tracheal phlegmon impact intensive care stay, hospital stay, mortality, and Health-related quality of life?

Participants will be followed up after undergoing tracheostomy for 7 days to identify eventual phlegmons.

At the two-year follow-up, the health-related quality of life will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Presence of indication for tracheostomy

Exclusion Criteria:

* Failure of the percutaneous tracheostomy technique or recourse to surgical tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Intensive Care undergoing percutaneous tracheostomy for any cause
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Neck phlegmon | 7 days
  Neck phlegmon in the incisional site

SECONDARY OUTCOMES:
Intensive Care Stay | 1 year
  Days of ICU stay
Hospital Stay | 1 year
  Days of hospital stay
Mortality | 30 days
  30 days mortality
Health related quality of life | 2 years
  15D instrument
Dysphagia | 2 years
  Eating Attitude test - EAT-10 questionnaire
Dysphonia | 2 years
  Voice Handicap Index - VHI-10 questionnaire
Dyspnoea | 2 years
  Modified Medical Research Council Dyspnea Scale - mMRC-10
Cough | 2 years
  Leicester Cough Questionnaire - LCQ

CONTACTS AND LOCATIONS:
Locations (1):
- Maggiore Hospital Carlo Alberto Pizzardi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Silvester W, Goldsmith D, Uchino S, Bellomo R, Knight S, Seevanayagam S, Brazzale D, McMahon M, Buckmaster J, Hart GK, Opdam H, Pierce RJ, Gutteridge GA. Percutaneous versus surgical tracheostomy: A randomized controlled study with long-term follow-up. Crit Care Med. 2006 Aug;34(8):2145-52. doi: 10.1097/01.CCM.0000229882.09677.FD. PMID 16775568
- [Background] Schindler A, Mozzanica F, Monzani A, Ceriani E, Atac M, Jukic-Peladic N, Venturini C, Orlandoni P. Reliability and validity of the Italian Eating Assessment Tool. Ann Otol Rhinol Laryngol. 2013 Nov;122(11):717-24. doi: 10.1177/000348941312201109. PMID 24358633
- [Background] Forti S, Amico M, Zambarbieri A, Ciabatta A, Assi C, Pignataro L, Cantarella G. Validation of the Italian Voice Handicap Index-10. J Voice. 2014 Mar;28(2):263.e17-263.e22. doi: 10.1016/j.jvoice.2013.07.013. Epub 2013 Oct 2. PMID 24094800
- [Background] Sorano A, Fumagalli C, Cinelli E, Birring SS, Fontana GA, Lavorini F. Development of an Italian version of the Leicester cough questionnaire and its relationship with other symptom-specific measures for patients with chronic cough. Respir Med. 2024 Jun;227:107642. doi: 10.1016/j.rmed.2024.107642. Epub 2024 Apr 24. PMID 38670318
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. PLoS Med. 2007 Oct 16;4(10):e296. doi: 10.1371/journal.pmed.0040296. PMID 17941714
- [Result] Mehta AK, Chamyal PC. TRACHEOSTOMY COMPLICATIONS AND THEIR MANAGEMENT. Med J Armed Forces India. 1999 Jul;55(3):197-200. doi: 10.1016/S0377-1237(17)30440-9. Epub 2017 Jun 26. PMID 28775631
- [Result] Voelker MT, Wiechmann M, Dietz A, Laudi S, Bercker S. Two-Year Follow-Up After Percutaneous Dilatational Tracheostomy in a Surgical ICU. Respir Care. 2017 Jul;62(7):963-969. doi: 10.4187/respcare.05290. Epub 2017 May 2. PMID 28465381